CLINICAL TRIAL: NCT03290131
Title: A Randomized, Double-Blind, Placebo-Controlled Parallel Group Study to Investigate the Safety and Efficacy of Arbaclofen Extended-Release Tablets for the Treatment of Spasticity in Patients With Multiple Sclerosis
Brief Title: A Study to Investigate the Safety and Effectiveness of Arbaclofen Extended-Release Tablets for Patients With MS
Acronym: OS440-3004
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: RVL Pharmaceuticals, Inc. (Industry)
Collaborators: Osmotica Pharmaceutical US LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: OS440-3004
Record Dates: First submitted 2017-09-19; First posted 2017-09-21 (Actual); Results first posted 2022-07-15 (Actual); Last update posted 2022-07-15 (Actual); Status verified 2022-05

CONDITIONS: Multiple Sclerosis; Spasticity, Muscle
MeSH Terms: conditions — Multiple Sclerosis; Muscle Spasticity | interventions — arbaclofen placarbil

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- AERT 40 mg (Active Comparator): 40 mg Arbaclofen Extended-Release Tablets
  Interventions: Drug: Arbaclofen
- AERT 80 mg (Active Comparator): 80 mg Arbaclofen Extended-Release Tablets
  Interventions: Drug: Arbaclofen
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Arbaclofen — Arbaclofen Extended Release Tablet
  Other Names: AERT
  Arms: AERT 40 mg; AERT 80 mg
Drug: Placebo — Placebo comparator
  Arms: Placebo

SUMMARY:
Multiple Sclerosis (MS) is an acquired inflammatory demyelinating disease of the central nervous system (CNS) that is regarded as the foremost cause of non-traumatic neurologic disability in adults in North America. Spasticity is a common complication in MS and occurs in up to 84% of patients. The main sign of spasticity is resistance to passive limb movement characterized by increased resistance to stretching, clonus, and exaggerated deep reflexes. Osmotica Pharmaceutical is currently developing arbaclofen extended-release tablets (AERT) for the treatment of spasticity in patients with MS.

DETAILED DESCRIPTION:
This is a multicenter, randomized, double-blind, placebo-controlled, parallel-group study to evaluate the safety and efficacy of oral AERT in MS patients with spasticity. Two doses of AERT, 40 mg and 80 mg, will be compared with placebo. The treatment groups will be randomized in a 1:1:1 ratio. Eligible patients will undergo a washout period for withdrawal of all medications used for anti-spasticity and/or muscle relaxation prior to randomization. A baseline clinical evaluation will be performed (Visit 2) to confirm eligibility for study randomization, and subjects will be randomly assigned to 1 of 3 treatment arms. Subjects will remain on maintenance treatment for approximately 3 months.

ELIGIBILITY:
Inclusion Criteria Includes:

* Subjects 18 to 65 years of age, inclusive.
* An established diagnosis of MS that manifests a documented history of spasticity.
* If receiving disease-modifying medications (eg, interferons approved for MS, glatiramer acetate, natalizumab, fingolimod, or mitoxantrone), there must be no change in dose for at least 3 months prior to Visit 1 (Screening), and the subject must be willing to maintain this treatment dose for the duration of the study. If receiving AMPYRA® (dalfampridine, fampridine, 4-amino puridine), subject must be at a stable dose for at least 3 months prior to Visit 1.
* Stable regimen for at least 3 months prior to Visit 2 for all medications and non-pharmacological therapies that are intended to alleviate spasticity.
* Absence of infections, peripheral vascular disease, painful contractures, advanced arthritis, or other conditions that hinder evaluation of joint movement.
* Use of a medically highly effective form of birth control (see Section 7.8) during the study and for 3 months thereafter for women of child-bearing potential (including female subjects and female partners of non-sterile male subjects).
* Willing to sign the informed consent form (ICF).

Exclusion Criteria Includes:

* Any concomitant disease or disorder that has symptoms of spasticity or that may influence the subject's level of spasticity.
* Concomitant use of medications that would potentially interfere with the actions of the study medication or outcome variables.
* Pregnancy, lactation, or planned pregnancy during the course of the study and for 3 months after the final study visit.
* Subject has clinically significant abnormal laboratory values, in the opinion of the investigator, at Visit 1 or Visit 2.
* Current malignancy or history of malignancy that has not been in remission for more than 5 years, except effectively treated basal cell skin carcinoma.
* Any other significant disease, disorder, or significant laboratory finding which, in the opinion of the investigator, puts the subject at risk because of participation, influences the result of the study, or affects the subject's ability to participate.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 536 (Actual)
Dates: Start 2018-01-28 (Actual); Primary Completion 2018-12-03 (Actual); Study Completion 2019-01-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Jacobs, MD, Study Director — Vice President
Locations (30):
- Belarus (5):
  - Grodno Regional Clinical Hospital, Grodno
  - Minsk City Clinical Hospital #5, Minsk
  - Minsk Scientific and Practical Center of Surgery, Transplantology and Hematology, Minsk
  - Republican Research and Development Center for Neurology and Neurosurgery, Minsk
  - Vitebsk Regional Diagnostic Center, Vitebsk
- Bosnia and Herzegovina (2):
  - University Clinical Centre of the Republic of Srpska, Clinic of Neurology, Banja Luka
  - University Clinical Hospital Mostar, Clinic of Neurology, Mostar
- Bulgaria (6):
  - Multiprofile Hospital for Active Treatment - Pleven within the structure of Military Medical Academy, Sofia, Pleven
  - University Multiprofile Hospital for Active Treatment "Dr. Georgi Stranski", Pleven, Clinic of Neurological Diseases, Pleven
  - Medical Center "Rusemed" EOOD, Rousse
  - Multiprofile Hospital for Active Treatment "ACIBADEM City Clinic Tokuda Hospital", Sofia, Neurology and Sleep Medicine Clinic, Sofia
  - Multiprofile Hospital for Active Treatment of Neurology and Psychiatry "Sveti Naum", Sofia, Sofia
  - University Multiprofile Hospital for Active Treatment "Sveti Ivan Rilski", Sofia, Clinic of Neurology Diseases, Sofia
- Croatia (4):
  - Clinical Hospital Center Osijek, Clinic of Neurology, Osijek
  - Clinical Hospital Center Rijeka, Department of Neurology, Rijeka
  - General Hospital Varazdin, Department of Neurology, Varaždin
  - Clinical Hospital Dubrava, Department of Neurology, Zagreb
- Moldova (2):
  - Institute for Emergency Medicine, Chisinau
  - National Institute of Neurology and Neurosurgery, Chisinau
- Poland (7):
  - Dendryt Medical Center, Katowice
  - Neuro-Medic, Katowice
  - Neurology Center Krzysztof Selmaj, Lodz
  - Medical Practice Professor K. Rejdak, Lublin
  - MED-Polonia, Sp. z o.o. (LLC), Poznan
  - "MEDYK" Stanislaw Mazur Sp. z o.o. (LLC) Medical Centre, Rzeszów
  - NeuroProtect Medical Center, Warsaw
- Serbia (4):
  - Clinical Center of Serbia, Belgrade
  - Clinical Hospital Center Zemun, Department of Neurology, Belgrade
  - Clinical Hospital Center Zvezdara, Belgrade
  - Clinical Center Kragujevac, Kragujevac

RESULTS

PARTICIPANT FLOW:
Groups:
- AERT 40 mg: 40 mg//day Arbaclofen Extended-Release Tablets
- AERT 80 mg: 80 mg/day Arbaclofen Extended-Release Tablets
- Placebo: Placebo Tablets
Period: Overall Study
Arm/Group | AERT 40 mg | AERT 80 mg | Placebo
Started | 179 | 179 | 178
Completed | 137 | 107 | 159
Not Completed | 42 | 72 | 19
Not completed — Adverse Event | 22 | 57 | 11
Not completed — Withdrawal by Subject | 18 | 13 | 8
Not completed — MS Relapse | 2 | 1 | 0
Not completed — Unknown reason | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- AERT 40 mg: 40 mg/day Arbaclofen Extended-Release Tablets
- Total: Total of all reporting groups
Arm/Group | AERT 40 mg | AERT 80 mg | Placebo | Total
Number analyzed (Participants) | 179 | 179 | 178 | 536
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 179 | 179 | 178 | 536
  >=65 years | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 108 | 101 | 110 | 319
  Male | 71 | 78 | 68 | 217
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 0 | 1 | 3
  Not Hispanic or Latino | 169 | 172 | 171 | 512
  Unknown or Not Reported | 8 | 7 | 6 | 21
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 4 | 0 | 2 | 6
  White | 171 | 177 | 174 | 522
  More than one race | 1 | 0 | 1 | 2
  Unknown or Not Reported | 3 | 2 | 0 | 5
Total Numeric-Transformed Modified Ashworth Scale (Most Affected Limb) [Mean (Standard Deviation); unit: units on a scale] — Total Numeric-Transformed Modified Ashworth Scale (TNmAS) is a 6-point scale to measure abnormality in tone or the resistance to passive movements. Higher score is worse outcome.
  For each joint, the minimum score is 0; maximum score is 5. The values for each of the 3 main joints are summed for the limb score. The limb with the highest score is the most affected limb (MAL). The highest possible score for a limb is 15. Limb range: 0 to 15.
  To arrive at total limbs (TL) score the values for all 4 limbs are summed; maximum total limb score is 60. TL range: 0 to 60.
  units on a scale | 7.4 (3.24) | 7.6 (3.02) | 7.6 (3.13) | 7.5 (3.1)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Total Numeric-transformed Modified Ashworth Scale Score of the Most Affected Limb (TNmAS-MAL)
Description: Total Numeric-Transformed Modified Ashworth Scale (TNmAS) is a 6-point scale to measure abnormality in tone or the resistance to passive movements. Higher score is worse outcome.
  For each joint, the minimum score is 0; maximum score is 5. The values for each of the 3 main joints are summed for the limb score. The limb with the highest score is the most affected limb (MAL). The highest possible score for a limb is 15. Limb range: 0 to 15.
  To arrive at total limbs (TL) score the values for all 4 limbs are summed; maximum total limb score is 60. TL range: 0 to 60.
Time Frame: 84 days
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | AERT 40 mg | AERT 80 mg | Placebo
Number analyzed (Participants) | 179 | 179 | 178
units on a scale | -1.7 (1.97) | -2.0 (1.78) | -1.4 (1.82)

2. Primary Outcome: Clinical Global Impression of Change (CGIC)
Description: The Clinical Global Impression of Change (CGIC) was developed to provide a brief, stand-alone assessment of the clinician's view of the subject's global functioning prior to and after initiating a study medication. The scale ranges from -3 to +3 judging whether the change is significantly worse (-3) to significantly improved (+3). Higher score is better outcome. The CGIC scale will be used to measure the overall change in the subject's condition since starting the study. There is no baseline value because the score is a measure of how the patient changed from baseline (treatment initiation).
Time Frame: 84 days
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Placebo: Placebo Tablets
  P
Arm/Group | AERT 40 mg | AERT 80 mg | Placebo
Number analyzed (Participants) | 179 | 179 | 178
units on a scale | 0.6 (1.0) | 0.4 (1.23) | 0.6 (0.94)

ADVERSE EVENTS:
Time Frame: Adverse event data collected over 92 day period.
Arm/Group | AERT 40 mg | AERT 80 mg | Placebo
All-Cause Mortality (participants affected / at risk) | 0/179 | 0/179 | 0/178
Serious Adverse Events (participants affected / at risk) | 7/179 | 6/179 | 6/178
Other Adverse Events (participants affected / at risk) | 148/179 | 154/179 | 133/178
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AERT 40 mg (N=179) | AERT 80 mg (N=179) | Placebo (N=178)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Withdrawal Syndrome (General disorders) | 0 (0) | 0 (0) | 1 (1)
Urosepsis (Immune system disorders) | 0 (0) | 0 (0) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Hip Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Joint Injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Pneumothorax (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Schwannoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Multiple Sclerosis Relapse (Nervous system disorders) | 2 (2) | 3 (3) | 0 (0)
Restless Leg Syndrome (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Somnolence (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Status Epilepticus (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Trigeminal Neuralgia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Delirium (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Depression Suicidal (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Somatic Symptom Disorder (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Toxic Skin Eruption (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AERT 40 mg (N=179) | AERT 80 mg (N=179) | Placebo (N=178)
Urinary Tract Disorder (Renal and urinary disorders) | 56 (56) | 57 (57) | 67 (67)
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 43 (43) | 40 (40) | 27 (27)
Asthenia (General disorders) | 24 (24) | 37 (37) | 27 (27)
Dizziness (Nervous system disorders) | 27 (27) | 35 (35) | 20 (20)
Nausea (Gastrointestinal disorders) | 40 (40) | 30 (30) | 28 (28)
Somnolence (Nervous system disorders) | 20 (20) | 27 (27) | 19 (19)
Vomiting (Gastrointestinal disorders) | 14 (14) | 19 (19) | 16 (16)
Gait Disturbance (General disorders) | 2 (2) | 14 (14) | 6 (6)
Headache (Nervous system disorders) | 4 (4) | 6 (6) | 12 (12)
Fatigue (General disorders) | 4 (4) | 10 (10) | 7 (7)
Vertigo (Ear and labyrinth disorders) | 5 (5) | 9 (9) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (2):
  • Study Protocol (2017-11-09): https://cdn.clinicaltrials.gov/large-docs/31/NCT03290131/Prot_000.pdf
  • Statistical Analysis Plan (2019-01-28): https://cdn.clinicaltrials.gov/large-docs/31/NCT03290131/SAP_001.pdf